CLINICAL TRIAL: NCT02698852
Title: A Prospective, Multicenter Trial Program in China to Evaluate the Efficacy and Safety of BuMA Supreme (eG Grafting) Biodegradable Polymer Sirolimus Eluting Stent in Patients With de Novo Coronary Lesions, OPC Trial
Brief Title: A Study to Evaluate the Efficacy and Safety of BuMA Supreme Drug Eluting Stent(DES)
Acronym: OPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIONEER-II, OPC, P02
Record Dates: First submitted 2016-01-05; First posted 2016-03-04 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Drug eluting stents; Interventional Cardiology
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BuMA Supreme group (Experimental): Totally 1000 subjects combined the 220 subjects from randomized controlled trial(RCT) group
  Interventions: Device: BuMA Supreme

INTERVENTIONS:
Device: BuMA Supreme — Stent platform: cobalt-chromium alloy

SUMMARY:
PIONEER-II OPC trial is a prospective, multicenter, single-arm registry trial. 1000 subjects from approximately 40 interventional cardiology centers will be enrolled to evaluate the target lesion failure(TLF) as the primary endpoint at 1 year. And all the subjects will be followed up to 5 years to attain the data of the secondary endpoints.

DETAILED DESCRIPTION:
Realizing even more uniform and complete endothelial coverage, BuMA Supreme™ biodegradable drug coating coronary stent system comprises a new generation of biodegradable drug eluting stent under development by Sino medical science(SINOMED). BuMA Supreme™ reconfigures BuMA™ DES utilizing a high caliber cobalt chromium platform coated with rapidly degrading PLGA scaffold.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, male or non-pregnant female
2. Evidence of non-symptomatic ischemia, stable or non-stable angina pectoris or past MI
3. Target lesion is primary and de-novo coronary artery disease
4. The target lesion length ≤ 60 mm, diameter 2.25mm-5.0mm (visually estimated)
5. Lesion diameter stenosis ≥70% (visually estimated)
6. For each target lesion, same stent implantation only
7. Acceptable candidate for Coronary Artery Bypass Grafting(CABG)
8. Understand the study purpose, willing to participate and sign the letter of consent, agrees to the follow-up visits including a 9 month angiographic follow-up

Exclusion Criteria:

1. Acute MI within 1 week
2. Chronic total occlusion(TIMI 0), left main lesion, intervention-required three-vessel lesions, branch vessel diameter ≥ 2.5mm and bypass lesion
3. More than 3 stents required
4. Patients refuse to be implanted stent
5. Calcified lesion failed in pre-dilation, twisted lesion and lesion unsuitable for stent delivery and expansion
6. In-stent restenosis
7. Planned percutaneous coronary intervention (PCI) within 3 months post procedure
8. Other stents implanted within 1 year
9. Severe heart failure (NYHA above III) or left ventricle ejection fraction(EF) <40%
10. Renal function damage, blood creatinine > 176.82 μmol/L
11. Bleeding tendency, active peptic ulcer disease, cerebral or subarachnoid hemorrhage, cerebral apoplexy within half year and contraindication for any anti-platelet or anticoagulation agents
12. Allergic to drugs or agents used in stent or protocol (PLGA, sirolimus, aspirin, clopidogrel, contrast agent, cobalt, nickel, chromium, iron, wolfram et. al.)
13. Life expectation < 12 months
14. Have not reached the primary end point when participating in other trial
15. Poor compliance to the protocol
16. Heart implantation cases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure | 1 year
  Target Lesion Failure(TLF) is defined as cardiac death, target vessel myocardial infarction(MI), or clinically-driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Stent implantation success rate | 5 years after PCI
  The stent implantation success rate includes device, lesion and clinical success rate.
Device-oriented Composite Endpoint(DoCE) | 1, 6, 12 month, and annually up to 5 years post procedure
  Device-oriented Composite Endpoint is defined as cardiac death, target vessel MI, or clinically-driven TLR (TLF).
Patient-oriented Composite Endpoint (PoCE) | 1, 6, 12 month, and annually up to 5 years post procedure
  Patient-oriented Composite Endpoint is defined as all cause death, all MI, or any revascularization.
Academic Research Consortium(ARC) defined stent thrombosis | 5 years after PCI
  Definite and probable stent thrombosis during acute, subacute, later and very late phase.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Shanghai Zhongshan Hospital; Shubin Qiao, M.D., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Yundai Chen, M.D., Study Director — Chinese PLA General Hospital; Shaoping Nie, M.D., Study Director — Beijing Anzhen Hospital; Yawei Xu, M.D., Study Director — Shanghai 10th People's Hospital; Xiangqing Kong, M.D., Study Director — Jiangsu Proving Hospital; Lang Li, M.D., Study Director — First Affiliated Hospital of Guangxi Medical University; Xiangqian Shen, M.D., Study Director — Central South University; Hui Li, M.D., Study Director — Daqing oilfield general hospital; Linghong Shen, M.D., Study Director — Shanghai Chest Hospital; Xi Su, M.D., Study Director — Wuhan Asia Heart Hospital; Jiyan Chen, M.D., Study Director — Guangdong Provincial People's Hospital; Genshang Ma, M.D., Study Director — Zhongda Hospital; Xiaoshu Cheng, M.D., Study Director — Second Affiliated Hospital of Nanchang University; Guosheng Fu, M.D., Study Director — Run Run Shaw Hospital; Zesheng Xu, M.D., Study Director — Cangzhou Central Hospital; Bin Li, M.D., Study Director — Hainan General Hospital; Jianan Wang, M.D., Study Director — The Second Affiliated Hospital of Zhejiang University School of Medical College; Haichu Yu, M.D., Study Director — The Affiliated Hospital of Qingdao University; Guotai Shen, M.D., Study Director — Jiangxi Provincial People's Hopital; Xiandong Li, M.D., Study Director — Shengjing Hospital; Xianxian Zhao, M.D., Study Director — Changhai Hospital; Tingbo Jiang, M.D., Study Director — The First Affiliated Hospital of Soochow University; Mingzhe Li, M.D., Study Director — Xuzhou Central Hospital; Zheng Zhang, M.D., Study Director — LanZhou University; Bei Shi, M.D., Study Director — Zunyi Medical College; Jinyu Huang, M.D., Study Director — Affiliated Hangzhou First People's Hospital ,Zhengzhou University School of Medicine; Honghua Ye, M.D., Study Director — Hua Mei Hospital, University of Chinese Academy of Sciences(Ningbo No.2 Hospital); Guohai Su, M.D., Study Director — Jinan Central Hospital; Hanjun Pei, M.D., Study Director — The First Affiliated Hospital of BaoTou Medical College; Shaobin Jia, M.D., Study Director — General Hospital of Ningxia Medical University; Chun Liang, M.D., Study Director — Shanghai Changzheng Hospital; Ronghai Man, M.D., Study Director — Chifeng Municipal Hospital; Jinchuan Yan, M.D., Study Director — Affiliated Hospital of Jiangsu University; Xuchen Zhou, M.D., Study Director — The First Affiliated Hospital of Dalian Medical University; Zhenyu Yang, M.D., Study Director — Wuxi People's Hospital; Yuehui Yin, M.D., Study Director — The Second Affiliated Hospital of Chongqing Medical University; Chunlai Zeng, M.D., Study Director — The Central Hospital of Lishui City; Kejun Huang, M.D., Study Director — Henan Provincial Chest Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No